CLINICAL TRIAL: NCT05337397
Title: Outpatient Laser Ablation of Recurrent Non-muscle Invasive Bladder Cancer
Acronym: OPTIMA
Status: Recruiting | Type: Observational
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: OPTIMA
Record Dates: First submitted 2022-04-11; First posted 2022-04-20 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: Laser ablation
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prior pTa low grade Non-Muscle invasive bladder cancer: Patient with recurrent Pta low grade Non-Muscle invasive bladder cancer, with negative urine cytology, and tumor size between 1 and 3 cm.
  Interventions: Procedure: Laser ablation

INTERVENTIONS:
Procedure: Laser ablation — Laser ablation of non-Muscle invasive bladder tumors in outpatient settings.

SUMMARY:
Aim: To investigate the feasibility and tolerability of the Olympus Soltive laser in treatment of large recurrent low-grade Ta tumours in an outpatient setting.

Background: Non-muscle invasive bladder cancer (NMIBC) is associated with a high yearly recurrence rate up to to 61%. Patients affected are therefore referred to long-term or even life-long follow-up, which burdens both patients and health care system. Recurrent tumours are most frequently treated with TURBT followed by adjuvant intravesical treatment. Repeat TURBT includes a risk of morbidity from the procedure itself and from general anaesthetics, which the procedure requires. Patients with NMIBC are generally elderly, multi-morbid, and as a result, they often show a poor tolerability of general anaesthetics. Thus, the need for non-surgical treatment modalities is imminent and continuous investigations are performed in the field including active surveillance, chemoresection and device-assisted intravesical chemotherapy. Laser ablation is a technique gaining attention in the treatment of NMIBC, based on the prospects of an outpatient treatment modality, which could prove TURBT and general anaesthesia unnecessary in select patients.

Methods: The study will be conducted as a prospective feasibility study. Included patients will undergo outpatient laser ablation using the Olympus Soltive laser under local anaesthetics.

Patients will be included from Aarhus University Hospital (Denmark), Fundació Puigvert (Spain), Motol University Hospital (Czech Republic) and Institut Universitaire du Cancer Toulouse Oncopole (France).

Data will be reported to the eCRF in the online REDCap web application. The eCRF is stored on a secure server under the responsibility of the Department of Clinical medicine at Aarhus University in Denmark.

REDCap is a secure web application for building and managing online surveys and databases. The Database will be in agreement with the laws and regulations of the Danish Data Protection Agency and EU regulations (GDPR).

The sponsor will be overall responsible for the data entry in the eCRF, and the validity of the data collected at the specific sites. Each participant will be coded with a unique patient identifier to ensure pseudo anonymity.

Perspectives: This study will be the first multinational study with focus on feasibility of outpatient laser ablation of large bladder tumours between 1-3 cm. Outpatient laser ablation of these large tumours has the potential to reduce the number of TURBTs per patient, thus easing the life of patients with non-muscle invasive bladder cancer, with fewer surgical procedures as well as reducing the overall treatment related costs for society. If thulium laser ablation proves effective, the treatment modality would be easily implemented and available based on the small size of the machinery.

DETAILED DESCRIPTION:
The participant will be informed that they can at any time withdraw their consent without influence on their further treatment. Withdrawal can be both with regards to further recordings of data but also deletion of collected data upon request. In case of withdrawal of consent before surgery, the patient will be treated according to local guidelines and excluded from the study.

The consent form will be approved by The Regional Committees on Health Research Ethics. The investigators are obligated to ensure, that comprehensive information is provided orally and in writing to the participant.

In the case of new relevant information or the design of the study is significantly changed, the participants will be informed, and the consent form updated.

Study participants will be informed that a signed consent form grants national investigator approved project staff, direct access to study data and patient's health records. The consent form also allows inspectors from the respective national health authorities access, if requested, in order to allow the authorities to perform controls and checks.

Data management:

The study will comply with The General Data Protection Regulation and The Data Protection Act.

All data are kept confidential in a pseudo anonymized form, according to the GDPR and the Danish Data Protection Agency's guidelines. The investigators, who will code each participant enrolled in the study with a unique patient identification number, will assure this.

Information obtained on the participants is confidential and may only be disclosed if permitted by the participant through a signed consent form. The signed consent allows both sponsor, relevant investigators from the study and authorities to enter the patient file.

The data generated by the study will be available for inspection upon request by the representatives of the national and local health authorities.

ELIGIBILITY:
Inclusion Criteria:

* At least one tumour with a diameter > 1 cm
* Papillary/non-solid tumours
* Previous low-grade NMIBC
* Ability to understand the participant information orally and in writing, in Danish, Spanish, Czech or French respectively
* Signed consent form

Exclusion Criteria:

* Tumour diameter > 3cm
* Tumour in the prostatic urethra
* Previous CIS, high-grade disease or muscle invasive bladder cancer with no later low-grade recurrence
* Positive cytology within 3 months (testing not mandatory in patients with low-grade tumours)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the follow up programme for Non-Muscle invasive Bladder Cancer in accordance with the European guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Succesful laser ablations | 4 months
  The proportion of successful laser ablation outpatient procedures compared to failed procedures leading to standard TURBT

SECONDARY OUTCOMES:
VAS score | day 0
  Pain during procedure, from 0(no pain) to highest pain(10)

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen B Jensen, Professor, MD, Principal Investigator — Skejby University Hospital: Aarhus Universitetshospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No